CLINICAL TRIAL: NCT03640416
Title: The Feasibility to Use Wearable Devices to Collect Physiologic Data During Night Shifts - A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0375-17-RMB
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Sleep Deprivation; Stress
Keywords: night on call; sleep deprivation; fitbit®; smart watch; stress
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Masking Description: No masking needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical residents (Other): Rambam Health Care Campus medical residents who work nights on call. Fitbit® Charge HR smart watch
  Interventions: Device: Fitbit® Charge HR smart watch

INTERVENTIONS:
Device: Fitbit® Charge HR smart watch — The Fitbit® Charge HR is a commercial product widely used worldwide, and data from the device is sent to a secured online server and can be accessed by each user to see only data collected from his own device. Data collected from the Fitbit® Charge HR is described earlier.

SUMMARY:
There is an increase interest in the use of wearable activity trackers and wearable technology in the various medical fields. Such devices can increase physical activity and decrease weight significantly.

Field and laboratory studies have shown that shift work can alter circadian rhythms, disrupt the sleep cycle, and hinder human performance. Sleep deprivation reduces alertness level, and may increase reaction time, cause memory impairment and impaired motor skills. Disrupted circadian rhythms, a well-known consequence of atypical work schedules, have been linked to neurodegeneration.

The aim of this pilot study is to evaluate the feasibility of wearable devices to collect data on physiologic parameters during sleep and awake under stress conditions.

The study population will include 30 Rambam Health Care Campus medical residents who work nights on call. The length of experiment per participant will be one month.

Subjective data on stress will be collected during the study. Data on vital signs and sleep stages will be collected through a smart watch Fitbit® Charge HR.

DETAILED DESCRIPTION:
Background There is an increase interest in the use of wearable activity trackers and wearable technology in the various medical fields. Such devices can increase physical activity and decrease weight significantly.

Shift work is usually referred to as dividing working hours among two or more occupational groups in order to cover the time needed for duty performance or for production process, and shift workers perform duties outside the regular working hours.

Field and laboratory studies have shown that shift work can alter circadian rhythms, disrupt the sleep cycle, and hinder human performance. Sleep deprivation reduces alertness level, and may increase reaction time, cause memory impairment and impaired motor skills. Disrupted circadian rhythms, a well-known consequence of atypical work schedules, have been linked to neurodegeneration.

Aim:

A pilot study to evaluate the feasibility of wearable devices to collect data on physiologic parameters during sleep and awake under stress conditions (night shifts).

Secondary objective: To assess physiological parameters collected by wearable devices. This study will help us assess the contribution of wearable devices to collect Big Data for future clinical studies.

Study design:

This is a prospective pilot study. The study population will include 30 Rambam Health Care Campus medical residents who work nights on call (not restricted to emergency departments).

A mobile phone application has been developed for the study. The application will be installed on each participant's smart phone (with Android operating system), and it will collect data on number of calls and SMS received during a night on call.

The participant will register to the mobile application without the need for a mobile number or e-mail address. The data collected will not be linked to a phone number or other personal information. Only the investigators of the Pediatric Pulmonology institute will have access to the data collected by the mobile application.

Only the data on number of calls and SMS will be collected during a night on call. The data will not include the content of the calls or SMS or the phone number of the sender or receiver of the calls and SMS.

Vital signs and data on sleep quality will be collected through a wearable device, which interacts with the mobile application. The wearable device used will be the Fitbit® Charge HR. Recent studies have shown that this wearable device provides an accurate measurement of heart rate during walking and running activities and energy expenditure . The device has been shown to have high accuracy in sleep evaluation and circadian rest-activity rhythm measurement (8.

The Fitbit® Charge HR collects data on:

* Continuous heart rate monitoring (heart beats per minute (BPM), average resting heart rate, and time spent in heart-rate zones)
* Sleep stages (light, deep and REM [Rapid Eye Movement) sleep) and auto sleep tracking
* Periods of time stationary vs. active (walked at least 250 steps)
* Steps taken
* Distance covered
* Calories burned The Fitbit® Charge HR is a commercial product widely used worldwide, and data from the device is sent to a secured online server and can be accessed by each user to see only data collected from his own device.

Each participant will provide written informed consent including:

1. Approval to join the experiment.
2. Information on Age, gender, height.
3. Telephone number.
4. Approval to collect time of SMS and phone calls.
5. Approval to provide all data collected from the wearable device.
6. Approval to collect hair and blood sample. It should be emphasized that all data on each participant will be collected anonymously, and no data will be provided to the health management of Rambam or any 3rd party.

Each participant will be given a coded name (starting STR1, STR2 etc..), and only the principal investigator will have access to the real name and ID numbers of the participants In addition, no genetic testing will be performed on hair or blood samples.

Visit 1 - recruitment

At the beginning of the experiment, each participant will schedule a at 9-10 am with an investigator in which the participant will:

* receive detailed information about the study, including data collection, privacy and security issues.
* sign an informed consent form.
* provide a table of nights on call for the month of the experiment.
* receive the activity wearable device and instructions on its functionality and requirements.
* provide demographic information.
* Assess baseline stress level:

  * Provide a hair sample (0.5 gr) for cortisol measurements.
  * Complete PSS - Perceived Stress Scale questionnaire (12).
  * Provide a blood test (6 ml) to evaluate stress hormones and specific cytokines for assessing stress. The serums will be stored and for any future use an amendment will be submitted to the Rambam helsinky committee.
  * Digit-span test - measures working memory's number storage capacity. The participant hears a sequence of numerical digits and is asked to recall the sequence correctly, with increasingly longer sequences being tested in each trial. The participant's span is the longest number of sequential digits that can accurately be remembered.
  * PASAT - Paced Auditory Serial Addition Test - measures capacity and rate of information processing and sustained and divided attention. The participant is given a number every 3 seconds and is asked to add the number he just heard with the number he heard before.

Trail Making test - cellular application that provides information about visual search speed, scanning, The test consists of two parts: in the first, the targets are all numbers (1, 2, 3, etc.) and the test taker needs to connect them in sequential order; in the second part, the subject alternates between numbers and letters (1, A, 2, B, etc.).

Data collection during month of participation:

Around each night on call of a participant:

1. From 24 hours before the night on call: Charge and wear the wearable. It is preferred that participants wear the device continuously throughout the month, except when charging.
2. During the night on call:

   * Continuous tracking of vitals, steps, sleep time and quality will be recorded.
   * 1-4 SMS messages will be sent randomly by one of the investigators of the Pediatric Pulmonology institute asking the participant to send a number between 1 and 5 indicating their subjective stress (1 means no stress and 5 means very stressed). Data will be collected by the investigator, no data will be saved on a remote server.
3. From night on call end until 24 hours later: continue wearing the wearable device.
4. 24 hours after the end of night on call (10:00 in the morning): respond to a message from one of the investigators to provide subjective stress level.

   Visit 2:
5. Immediately after one of the nights on call (9:00-10:00 in the morning):

   1. Participants will complete a second PSS - Perceived Stress Scale questionnaire (9).
   2. Blood pressure and heart rate will be measured.
   3. a 5 ml blood sample will be collected.
   4. Digit-span test, PASAT, Trail Making test will be preform again The visits will be scheduled and done in the Rambam health care campus in a location and timing suitable to the participant.

Data analysis After data collection, we will build a statistical model that will try to estimate stress based on behavioral characteristics.

Stress will be estimated using:

1. Self-reports (scale of 1-5 on subjective stress through random messages from the study mobile application during night on call).
2. Heart rate, heart rate variability, blood pressure.
3. Digit-span test, PASAT, Trail Making test before and after nightshift will be analyzed 3 Digit-span test, PASAT, Trail Making test will be preform again The behavioral characteristics will include:

1. Length and time of sleep before, during and after a shift, and sleep stages tracking (light, deep and REM sleep) 2. Interruptions (SMS, calls, movement) during wake and sleep 3. Movement during the shift (time while being stationary vs. active)

ELIGIBILITY:
Inclusion Criteria:

1. A medical resident working nights on call at Rambam.
2. Use a smart phone (Android OS) with a data plan.

Exclusion Criteria:

1. Pregnancy and lactation.
2. Medications:

   1. CNS (Central Nervous System) stimulants - Ritalin (methyphenidate), Concerta.
   2. Beta Blockers, Calcium channel Blockers
   3. glucocorticoids
   4. Sedatives
3. Unwilling to carry smart phone or wearable device on a continuous basis during shifts and at least 24 hours before and after shifts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
assessment of sleep duration (hours) | one month per participant
  calculated using the Fitbit® charge HR device

SECONDARY OUTCOMES:
heart rate (beats/mins) | one month per participant
  taken using the Fitbit® charge HR device
blood pressure (mmhg) | one month per participant
  measures during the night on call
steps taken (number) | one month per participant
  taken using the Fitbit® charge HR device
Trail Making test | one month per participant
  Trail Making test - cellular application that provides information about visual search speed, scanning, The test consists of two parts: in the first, the targets are all numbers (1, 2, 3, etc.) and the test taker needs to connect them in sequential order; in the second part, the subject alternates between numbers and letters (1, A, 2, B, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No